CLINICAL TRIAL: NCT03907475
Title: DURVA+ : Evaluation of the Safety and Pharmacodynamics of Anti-PD-L1 Antibody Durvalumab in Combination With Chemotherapy in Patients With Advanced Solid Tumors
Brief Title: Durvalumab in Combination With Chemotherapy in Treating Patients With Advanced Solid Tumors, DURVA+ Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01886; NCI-2019-01886 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10292 (Other: National Cancer Institute LAO); 10292 (Other: CTEP); ZIABC011078 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Capecitabine; Carboplatin; durvalumab; Immunoglobulin G; Disulfides; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm I (durvalumab) (Active Comparator): Patients receive durvalumab IV over 60 minutes on days 1 and 15 of cycles 1 and 2 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab
- Arm II (gemcitabine hydrochloride, durvalumab) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and durvalumab IV over 60 minutes on days 8 and 22 of cycles 1 and 2 and day 8 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who discontinue gemcitabine hydrochloride continue receiving durvalumab alone as in Arm I. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Gemcitabine Hydrochloride
- Arm III (pegylated liposomal doxorubicin, durvalumab) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and durvalumab IV over 60 minutes on days 8 and 22 of cycles 1 and 2 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Echocardiography Test; Drug: Pegylated Liposomal Doxorubicin Hydrochloride
- Arm IV (capecitabine, durvalumab) (Experimental): Patients receive capecitabine PO BID on days 1-14, and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Biological: Durvalumab
- Arm V (carboplatin, durvalumab) (Experimental): Patients receive carboplatin IV over 30-60 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Biological: Durvalumab
- Arm VI (paclitaxel, durvalumab) (Experimental): Patients receive paclitaxel IV over 60 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Paclitaxel
- Arm VII (nab-paclitaxel, durvalumab) (Experimental): Patients receive nab-paclitaxel IV over 30 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm IV (capecitabine, durvalumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm V (carboplatin, durvalumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Arm III (pegylated liposomal doxorubicin, durvalumab)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm II (gemcitabine hydrochloride, durvalumab)
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
  Arms: Arm VII (nab-paclitaxel, durvalumab)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm VI (paclitaxel, durvalumab)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Doxorubicin Liposomal; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm III (pegylated liposomal doxorubicin, durvalumab)

SUMMARY:
This phase II trial studies the side effects of durvalumab when given together with chemotherapy in treating patients with solid tumors that have spread to other places in the body (advanced). Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as gemcitabine hydrochloride, pegylated liposomal doxorubicin hydrochloride, capecitabine, carboplatin, paclitaxel, and nab-paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with durvalumab may improve how immune cells respond and attack tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of adding durvalumab to standard chemotherapy regimens.

SECONDARY OBJECTIVES:

I. Determine the changes that occur in the immune microenvironment in response to chemotherapy and assess how these changes alter the pharmacodynamic effects of a checkpoint inhibitor.

II. Investigate whether the response to immunotherapy correlates with patients' genetic aberrations and/or the activation status of tumor-infiltrating and circulating T cells.

III. Explore the relationship between immune status of the tumor and overall tumor mutational load.

IV. Assess preliminary antitumor activity of the durvalumab and chemotherapy combinations.

EXPLORATORY OBJECTIVE:

I. Assess whether changes in cell-free deoxyribonucleic acid (DNA) correlate with response or resistance to the study regimens.

OUTLINE: Patients are assigned to 1 of 7 arms.

ARM I: Patients receive durvalumab intravenously (IV) over 60 minutes on days 1 and 15 of cycles 1 and 2 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM II: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and durvalumab IV over 60 minutes on days 8 and 22 of cycles 1 and 2 and day 8 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who discontinue gemcitabine hydrochloride continue receiving durvalumab alone as in Arm I. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM III: Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and durvalumab IV over 60 minutes on days 8 and 22 of cycles 1 and 2 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) during screening. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM IV: Patients receive capecitabine orally (PO) twice daily (BID) on days 1-14, and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM V: Patients receive carboplatin IV over 30-60 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM VI: Patients receive paclitaxel IV over 60 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

ARM VII: Patients receive nab-paclitaxel IV over 30 minutes on day 1 and durvalumab IV over 60 minutes on day 8 of cycle 1, days 1 and 15 of cycle 2, day 8 of cycle 3, and day 1 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

After completion of study treatment, patients are followed up monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented metastatic or locally advanced (not amenable to surgery) solid tumors whose disease has progressed following at least one line of standard therapy and/or no standard of treatment exists that has been shown to prolong survival.

  * If anti-PD-1 or one of the 6 chemotherapy agents is standard-of-care, prior therapy with the agent would not be required.
* Patient must have tumor amenable to biopsy and be willing to undergo a tumor biopsy.

  * Flash frozen tissue collected as part of another study or from a procedure performed due to medical necessity may be acceptable as the baseline sample if the samples were collected within 3 months prior to registration and the patient has not received any investigational or targeted treatment since that time.
  * A patient who cannot be safely biopsied may be considered for the study upon discussion with Principal Investigator.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan.
* Patients with bone metastases or hypercalcemia on intravenous bisphosphonate treatment, denosumab, or similar agents are eligible to participate and may continue this treatment. Patients with prostate cancer may continue luteinizing hormone-releasing hormone (LHRH) agonists or antagonists.
* Age ≥ 18 years. Children are excluded from this study, but may be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Absolute neutrophil count >= 1,000/uL (mcL).
* Platelets >= 100,000/uL (mcL).
* Total bilirubin < 1.5 x institutional upper limit of normal.

  * This will not apply to patients with confirmed Gilbert syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only at the discretion of the principal investigator (PI), study chair or their designee.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal, or up to 5 x upper limit of normal (ULN) if liver metastases are present.
* Calculated creatinine clearance > 40 mL/min by the Cockcroft-Gault formula
* Any prior systemic therapy (including checkpoint inhibitors), or major surgery must have been completed >= 3 weeks (> 6 weeks for nitrosoureas or mitomycin C) or 5 half-lives of the agent, whichever is shorter, prior to enrollment on protocol, and toxicity from prior treatment must have recovered to eligibility levels. Radiation therapy must have been completed >= 1 week prior to starting treatment. Radiofrequency ablation (RFA) of localized lesions should have been performed >= 1 week prior to starting treatment. All radiation-related toxicity must have resolved to < grade 2.

  * Palliative radiotherapy is permitted between disease progression on Arm 1 and crossover to a combination therapy arm (Arms 2-7), provided there is a washout period of >= 1 week and any toxicity from radiation has resolved to < grade 2
  * Patients on any arm may receive palliative radiotherapy or loco-regional ablative therapy and remain on study, provided the radiation is not delivered to the target lesion and the patient does not have tumor progression by Response Evaluation Criteria in Solid Tumors (RECIST)
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon-alpha or interleukin-2) must have been completed at least 3 weeks before the first dose of durvalumab.
* Body weight > 30 kg.
* Human immunodeficiency virus (HIV)-infected (HIV1/2 antibody-positive) patients may participate if they meet all the following eligibility requirements:

  * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within the past 12 weeks.
  * They must have a CD4 count >= 250 cells/uL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/uL over the past 2 years, unless it was deemed related to chemotherapy-induced bone marrow suppression.

    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/uL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy.
  * They must have an undetectable viral load and a CD4 count >= 250 cells/uL within 28 days of enrollment.
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months.
  * Monitoring for HIV-infected patients should include:

    * Viral load and CD4 count every 8-10 weeks.
* The effects of targeted agents on the developing human fetus are unknown. The cytotoxic agents chosen for combination with durvalumab adversely affect human fertility and gestation. For these reasons, women of childbearing potential and men must agree to use highly effective contraception prior to study entry for the duration of study participation and for 6 months following the last dose of a study drug.
* Because there may be a risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued while the patient is on this trial and for 6 months following the last dose of study drug.
* Patients should be willing not to donate blood while participating in this study or for at least 90 days following the last dose of study drug.
* Left ventricular ejection fraction greater than 50% or the institutional lower limit of normal by echocardiography (ECHO) at entry (patients enrolling on Arm 3 only).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who received prior therapy with a checkpoint inhibitor and were taken off drug for serious adverse events are excluded. Patients who had prior CTLA-4 inhibitor treatment and did not experience serious adverse events are eligible for all arms. Patients who had prior PD-L1/PD-1 inhibitor treatment and did not experience serious adverse events are excluded from the durvalumab monotherapy arm but are eligible for the chemotherapy combinations.
* Patients with pancreatic cancer, prostate cancer, or microsatellite stable (MSS) colorectal cancer, or other histologies where clinical evidence exists that single-agent inhibition of PD-L1/PD-1 has minimal activity will not receive single-agent durvalumab but may be eligible to receive this agent with chemotherapy (Arms 2-7).
* Women who are pregnant or breastfeeding.
* Patients who are receiving any other investigational agents. Patients on other trials will be eligible as long as they are no longer receiving study treatment.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (e.g. bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. Patients with active tuberculosis (TB) are also excluded.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or glucocorticoid equivalent dose of another steroid
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Patients should not be vaccinated with live attenuated vaccines within 30 days before starting or after completing durvalumab treatment.
* Patients who have a history of seizures will not be eligible, unless they have either not had seizures or have been on stable doses of anti-seizure medicine and had no seizures for 4 weeks, in which case they will be eligible. Patients taking enzyme-inducing anticonvulsants (i.e., carbamazepine, fosphenytoin, oxcarbazepine, phenobarbital, phenytoin, primidone) will only be eligible for Arm 1 (durvalumab monotherapy) and Arm 2 (durvalumab + gemcitabine).
* Patients receiving warfarin are not eligible for Arm 4 (capecitabine) due to the potential for life-threatening interactions. Patients on warfarin are eligible to enroll in one of the other arms provided there is increased vigilance with respect to monitoring international normalized ratio (INR).
* Patients with uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the past 6 months, invasive fungal infections, or active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e., quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable HCV-ribonucleic acid [RNA]), are not eligible to participate. Testing for HBV-DNA and HCV-RNA will be mandatory for patients with hepatocellular carcinoma (HCC) only; testing for hepatitis B or other infections for eligibility will be performed only if clinically indicated.
* History of grade >= 2 infusion reactions or allergic reactions to humanized monoclonal antibodies. Exception: patients with a history of grade 2 infusion reactions to checkpoint inhibitors may be eligible if resumption of prior therapies with pre-medications has been documented without recurrence of infusion reactions of any grade; those patients should receive the same pre-medications with the first and subsequent doses of durvalumab.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 cycles (Arms 1-3) or 4 cycles Arms (4-7)

OTHER OUTCOMES:
Changes in the immune microenvironment | Baseline up to 3 months after the last dose of study drug
  Will assess how these changes alter the pharmacodynamic effects of a checkpoint inhibitor.
Immunotherapy response of tumor-infiltrating and circulating T cells | Up to 3 months after the last dose of study drug
  Will investigate whether the response to immunotherapy correlates with patients' genetic aberrations and/or the activation status of tumor-infiltrating and circulating T cells.
Immune status of the tumor and overall tumor mutational load | Up to 3 months after the last dose of study drug
  Will explore the relationship between immune status of the tumor and overall tumor mutational load.
Cell-free deoxyribonucleic acid (cfDNA) | On day 1 of each treatment cycle and at the time of disease progression
  Will be analyzed by MoCha with the TSO500 targeted sequencing assay (or similar assay) to quantitatively assess longitudinal changes (such as changes in circulating tumor DNA levels as a percentage of total circulating, cell-free DNA) and to identify any mutations that may be associated with study treatment sensitivity or resistance.

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (1):
- National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm